CLINICAL TRIAL: NCT07181278
Title: Optimization of HPV-based Cervical Cancer Screening Strategies Among Women Living With HIV: Effectiveness and Implementation of Decentralized Approach Using a Mobile Team With HPV Testing in the Western Region of Cameroon
Brief Title: Optimization of Cervical Cancer Screening Strategies Among Women Living With HIV: Effectiveness and Implementation of Decentralized Approach Using a Mobile Team With HPV Testing in the Western Region of Cameroon
Acronym: OptiTri_MT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Recherche pour le Developpement (Other Government)
Collaborators: International Agency for Research on Cancer (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Centre Pasteur du Cameroun (Other); Ecole Polytechnique Fédérale de Lausanne (Other); Queen Mary University of London (Other); Programme PACCI, Abidjan, Côte d'Ivoire (Unknown); RSD Institute, Cameroon (Unknown); Centre Hospitalier Simone VEIL de BEAUVAIS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: IRD_2024_CEPED_OptiTri_mobileT; 22SANIC204 (Other Grant/Funding Number: L'Initiative); ANRS 0467 (Other Grant/Funding Number: ANRS-MIE)
Record Dates: First submitted 2025-09-12; First posted 2025-09-18 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-09

CONDITIONS: Cervical Cancer Screening; HIV
Keywords: cervical cancer; screening; HIV; implementation; resource-limited setting; HPV test; decentralization; thermal ablation
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Mobile Health Units; Therapeutics

STUDY DESIGN:
Intervention Model Description: Stepped-wedge cluster randomized clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Centralized screening (Active Comparator): A self collected vaginal sample is collected onsite. All the other screening are performed in a reference centre.
  Interventions: Other: Centralized screening
- Decentralized arm (mobile team) (Experimental): A mobile team consisting of midwives and lab technician with a Genexpert platform visits the health centres and perform CC screening with HPV testing and treament when required.
  Interventions: Other: Mobile unit with quasi point of care HPV testing and immediate triage + treatment

INTERVENTIONS:
Other: Mobile unit with quasi point of care HPV testing and immediate triage + treatment — A mobile team consisting of one or two midwives and a lab technician with a Genexpert platform visits the health centres on a regular basis.
  After informed consent is granted, participants perform a vaginal self-sample, which is immediately analyzed with the Genexpert plateform. Participants who test HPV positive are invited for immediate triage and treatment if required.
  Arms: Decentralized arm (mobile team)
Other: Centralized screening — Self-collected samples are sent to a reference laboratory for HPV testing. Results are communicated to the participants and HPV positive women are invited to go to the reference centre where triage and treatment (when required) are performed.
  Arms: Centralized screening

SUMMARY:
Context. Cervical cancer (CC) is a leading cause of death among women living with HIV (WLHIV) in resource-limited settings. Yet, effective methods for screening and preventing CC are available. The recommanded approach for CC screening is based on multiple steps, including initial test to detect human papillomavirus (HPV) infection, visual inspection to identify women with HPV at risk for precancerous lesion and treatment when required.

Dropout may occur at these different steps, compromising the success of the CC elimination strategy. Performing all the screening and treatment sequences in a single visit has been recommanded based on the results of a large South African trial. Yet, in many contexts, including those with limited resources, the screening and treatment activities are performed in multiple visites for logistical reasons, resulting in many dropouts.

Different strategies for delivering screening with HPV testing for WLHIV are possible. A first approach ("centralized approach") consists of having well equipped reference centres with experienced health workers and referring women to these centers. An alternative consists of having a mobile unit who can bring equipment and health workers and perform the CC screening in the usual places of patient care ("decentralised" or mobile team approach). Each of these two approaches has advantages and limitations in terms of coverage, completeness, cost and quality of screening. It is necessary to evaluate them in real life to inform national decision-makers on the best strategy to use in their countries.

The OptiTri-MU study aims to evaluate and compare the effectiveness of these two strategies for delivering CC screening ("centralized" screening versus "decentralized" screening). It will also assess the implementation of each strategy and include three sub-studies designed to evaluate :

* the performance of urinary HPV testing.
* the performance of different methods to identify women requiring a treatment.
* the risk of post-treatment cervical disease. Design This is a trial in which the intervention (mobile team) will be implemented gradually. All sites starts with the centralized screening strategy. At each period, a new site is ransomly selected and start the the decentralized screening strategy. There will be 6 periods of 10 weeks. The effectiveness of the intervention will be assessed by comparing the outcomes at each site before and after implementation and by comparing the sites with each other. The primary outcome for effectiveness is the screening completeness 120 days after enrollment.

The study will also assess the implementation of each screening strategy in terms of :

* Success through the measure of fidelity, reach and completeness
* Identification of adaptation, barriers and facilitating/leverage factors
* Perception, feasibility and acceptability of the screening strategies (by patients and health care workers)

Other study objectives include :

* To assess the performance of different methods to identify women requiring a treatment
* To assess the performance of HPV testing on a urine sample compared with vaginal self-collected or cervical (clinician-collected) samples
* To assess the efficacy of treatment in terms of post-treatment cervical lesions Study population. Participants will be WLHIV aged 25 to 49 and eligible for CC screening. Health care workers will also be invited to participate to the implementation research. The data collected will be quantitative and qualitative.

DETAILED DESCRIPTION:
Context. Cervical cancer (CC) is a leading cause of death among women living with HIV (WLHIV) in resource-limited settings. Yet, effective methods for screening and preventing CC are available. The recommanded approach for CC screening is based on multiple steps, including initial test to detect human papillomavirus (HPV) infection, visual inspection to identify women with HPV at risk for precancerous lesion and treatment when required.

Dropout may occur at these different steps, compromising the success of the CC elimination strategy. Performing all the screening and treatment sequences in a single visit has been recommanded based on the results of a large South African trial. Yet, in many contexts, including those with limited resources, the screening and treatment activities are performed in multiple visites for logistical reasons, resulting in many dropouts.

Different strategies for delivering screening with HPV testing for WLHIV are possible. A first approach ("centralized approach") consists of having well equipped reference centres with experienced health workers and referring women to these centers. An alternative consists of having a mobile unit who can bring equipment and health workers and perform the CC screening in the usual places of patient care ("decentralised" or mobile team approach). Each of these two approaches has advantages and limitations in terms of coverage, completeness, cost and quality of screening. It is necessary to evaluate them in real life to inform national decision-makers on the best strategy to use in their countries.

The OptiTri-MU study aims to evaluate and compare the effectiveness of these two strategies for delivering CC screening ("centralized" screening versus "decentralized" screening). It will also assess the implementation of each strategy and include three sub-studies designed to evaluate :

* the performance of urinary HPV testing.
* the performance of different methods to identify women requiring a treatment.
* the risk of post-treatment cervical disease. Design It is a stepped-wedge cluster randomized trial with primary HIV care unit as clusters and 6 periods of 10 weeks. All sites starts with the centralized screening strategy. At each period, a new site is randomized to the decentralized screening strategy. The primary outcome for effectiveness is the screening completeness 120 days after enrollment.

The study will also assess the implementation of each screening strategy in terms of :

* Success through the measure of fidelity, reach and completeness
* Identification of adaptation, barriers and facilitating/leverage factors
* Perception, feasibility and acceptability of the screening strategies (by patients and health care workers)

Other study objectives include :

* To assess the performance of different methods to identify women requiring a treatment
* To assess the performance of HPV testing on a urine sample compared with vaginal self-collected or cervical (clinician-collected) samples
* To assess the efficacy of treatment in terms of post-treatment cervical lesions Study population. Participants will be WLHIV aged 25 to 49 and eligible for CC screening. Health care workers will also be invited to participate to the implementation research. The data collected will be quantitative and qualitative.

ELIGIBILITY:
Inclusion Criteria:

* Women
* HIV infection
* Age between 25 and 49 years old
* Receiving or starting ARV treatment
* Agreeing to participate in the study and having signed the consent

Exclusion Criteria:

* Current pregnancy
* Hysterectomy
* Treatment of cervical lesions within 12 months
* Expected follow-up difficulties: planned absence that could interfere with the participation in the study (e.g., travel abroad, relocation, imminent transfer, etc.);
* Any pathology or concomitant treatment which, in the opinion of the investigators, contraindicates participation or prevents satisfactory participation in the study

Deferred inclusion if

* menstrual bleeding
* Postpartum (<12 weeks after delivery)
* Clinical signs of cervical or pelvic infection

Ages: 25 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1180 (Estimated)
Dates: Start 2025-04-28 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Screening completeness | 120 days post screening initiation
  Proportion of HPV+ participants completing all screening steps within 60 days of inclusion.

SECONDARY OUTCOMES:
Screening completeness 2 | 60 days post screening initiation
  Proportion of HPV+ participants completing all screening steps within 60 days of inclusion.
Acceptability of the screening delivery strategy | Baseline (screening)
  Questionnaire assessing the acceptability and using a 4 point Likert scale
Triage performance | Baseline (screening)
  Sensitivity, specificity of the triage option to detect CIN2+ and CIN3+ lesion
Performance of urinary HPV test | Baseline (screening)
  Concordance between HPV test results from urine samples and those from cervical specimen collected by the clinician
Post treatment cervical lesion | 12 months post screening
  Frequency of CIN2+ lesion 12 months after treatment and performance of the markers of cure (sensitivity and specificity)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Debeaudrap, MD, PhD, Study Director — Institut de Recherche pour le Développement (IRD); Joëlle Sobngwi, MD, PhD, Principal Investigator — RSD Institute
Locations (6):
- Cameroon (6):
  - Bafoussam Baptist Hospital, Bafoussam
  - Bingo Hospital, Bafoussam
  - Centre Médical Spécialisé ACHA, Bafoussam
  - Hôpital Régional Annexe, Bafoussam
  - Bandjoun District Hospital, Bandjoun
  - Foumbot District Hospital, Foumbot

IPD SHARING:
Plan to Share IPD: No